## National Taipei University of Nursing and Health Sciences Doctoral Dissertation Proposal

## **School of Nursing**

The Effect of a Yoga Intervention for Reducing Stress among People Living
with HIV in Indonesia: A Randomized Controlled Trial
(Participant Informed Consent)

Jufri Hidayat

Advisor: Miao-Yen Chen RN, PhD

NCT Number: NCT05503680

Document date: January 7th, 20223

## Participant consent form



No. 365, Mingde Rd, Beitou District, Taipei City, 112, Taiwan

## **Participant Consent Form**

| Tittle project: | The effect of a yoga intervention for reducing stress among people living |
|---|---|
| | with HIV during covid-19 pandemic in Indonesia, a randomized |
| | controlled trial. |
| Student researcher: | Dr. (Cand) Jufri Hidayat RN, MScN |
| Supervisor: | Miao-Yen Chen RN, PhD |
| Ι | (the participant) have read and understood the information explained by |
| the researcher. Any question I asked, have been answered to my satisfaction | |

- Participate in this study which will last two months in total

I agree to:

- Complete baseline assessment questionnaires, then take the surveys again after eight
  weeks of yoga sessions, and finally, one more time a month after the yoga sessions are
  done.
- Complete the CD4 count or viral load test at baseline, again after finishing the eight-week yoga sessions, and one more time a month after the sessions are done.
- Participate in a home-based yoga intervention program via Zoom (every Thursday and Sunday afternoon at 3:00 pm).
- Give permission to the researcher to access my medical records.

I realize I can withdraw my consent at any time if it is not convenient for me to continue, without comment or penalty. I agree that research data collected for this study may be published or may be provided to other researchers in a form that does not identify me in any way.

| Name of participant | |
|----------------------------|---------|
| Signature | Date: |
| Name of student researcher | |
| Signature | . Date: |
| Name of supervisor | |
| Signature | Date: |